CLINICAL TRIAL: NCT04645563
Title: Using Whatsapp for the Consultation of Covid-19 Suspected Patients in Pandemic Polyclinics; A Retrospective Case Control Study
Brief Title: Using Whatsapp for the Consultation
Status: Completed | Type: Observational
Sponsor: Kafkas University (Other)
Responsible Party: Principal Investigator, Ramazan Sbirli, Dr., Kafkas University
Other Study IDs: Clinical-3
Record Dates: First submitted 2020-11-20; First posted 2020-11-27 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Covid-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Whatsapp Group: This group includes 54 patients who have consulted via whatsapp. The ID physician will be consulted for all the subjects once laboratory results and CT reports were complete. All the consultations were performed with the same smartphone, and every Whatsapp consultation held since the very beginning of the pandemic was evaluated.
  In this type of consultation, Thorax CT images of the patient were turned into a video of approximately 30-35 seconds, and during this video recording, the patient's clinical condition and laboratory results were also transferred to the ID physician. The ID physician, on the other hand, will state his/her admission-discharge decision via Whatsapp as "hospitalization" or "discharge". Eventually the consultation result will be recorded in the patient's folder. The moment the video was sent will be recorded as the beginning of the patient's consultation period and response time to whatsapp video will be saved as consultation response time.
  Interventions: Other: Sending thorax ct video images via smartphone applications
- Bedside Consultation Group: This group includes 90 patients who have consulted bedside. The patients that has problems which are concerning multiple consultation will be excluded.
  The ED physician wrote a consultation note over the hospital information system by specifying the patient's clinical status, history and laboratory parameters. A physician will be consulted for all the eligible subjects after their laboratory results and CT reports were complete. The ID physician examined the subjects at the bedside within 30 minutes (the legal response time in Turkey) of seeing the consultation request. Consultation response time will be saved as time between entering consultation information through the system to completion of the consultation note Although the consultant ID physicians will be informed via Whatsapp, they held the consultation at the bedside for the subjects they deemed appropriate.

INTERVENTIONS:
Other: Sending thorax ct video images via smartphone applications — Video images of the patients will be sent via smartphone application to infectious disease specialist for consulting.
  Groups: Whatsapp Group

SUMMARY:
Telephone, internet-connected devices (phablet, pc), chat platforms, mobile applications (Skype, Facebook messenger, Whatsapp, to name a few) can be exploited for telemedicine applications. Whatsapp and similar applications are widely used to facilitate clinical communication between physicians, too. Moreover, Whatsapp is used between ED physicians and consultant physicians during ED consultations in which medical information is exchanged. This platform is regarded as a useful application in the consultation of dermatological and orthopaedic cases. Preventing the overcrowding in the ED is key to reducing the transmission risk, and teleconsulting practice is thought to be effective in the diagnosis, treatment and reduction of the risk of disease transmission, most notably in the Covid-19 pandemic process. Video consulting is highly recommended in some countries on the grounds that it is likely to reduce the risk of transmission. Whatsapp-like applications are one of the video-consulting platforms assumed to reduce the risk of contamination by minimizing the patient-doctor contact.

This study thus sets out to investigate the effect of Whatsapp video consultation upon patient admission and discharge times in comparison to bedside consultation in the evaluation of potential Covid-19 patients visiting the Covid-19 outpatient clinic during the pandemic period.

The subjects who presented to ED Covid-19 outpatient clinic between March 11, 2020 and May 31, 2020 and for whom an infectious diseases (ID) physician was consulted (via Whatsapp or at bedside) will be included in the study in accordance with the inclusion and exclusion criteria. Eventually, 54 patients whose consultations were made via Whatsapp and 90 patients whose consultations were made at bedside will be in this study.

DETAILED DESCRIPTION:
Telephone, internet-connected devices (phablet, pc), chat platforms, mobile applications (Skype, Facebook messenger, Whatsapp, to name a few) can be exploited for telemedicine applications. Whatsapp and similar applications are widely used to facilitate clinical communication between physicians, too. Moreover, Whatsapp is used between ED physicians and consultant physicians during ED consultations in which medical information is exchanged. This platform is regarded as a useful application in the consultation of dermatological and orthopaedic cases. Preventing the overcrowding in the ED is key to reducing the transmission risk, and teleconsulting practice is thought to be effective in the diagnosis, treatment and reduction of the risk of disease transmission, most notably in the Covid-19 pandemic process. Video consulting is highly recommended in some countries on the grounds that it is likely to reduce the risk of transmission. Whatsapp-like applications are one of the video-consulting platforms assumed to reduce the risk of contamination by minimizing the patient-doctor contact.

Even though some studies on Whatsapp consultation in ED exist in the literature, we did not encounter any study investigating the effect of Whatsapp-mediated consultation on pandemic polyclinics.

This study thus sets out to investigate the effect of Whatsapp video consultation upon patient admission and discharge times in comparison to bedside consultation in the evaluation of potential Covid-19 patients visiting the Covid-19 outpatient clinic during the pandemic period.

During the coronavirus pandemic process, the patients were consulted with the ID department through the bedside consultation method or video transmission from Whatsapp. The consultation method of the patients will be scanned retrospectively (from the fixed ED phone and the hospital system) and will be recorded in the dataset. The method of consultation through video transmission will be implemented at the beginning of the pandemic process to increase communication between the emergency service and the infectious diseases department.

Duration of video that send on whatsapp for consultation, infection diseases specialist response to video, clinician's response to bedside consultation was saved to dataset. Besides, time from patients application to CT, time from patients application to lab results, duration of patients in emergency service, and time periods of consultation (within working hour [8:00-17:00], or out of working hours [17:00-08:00]) will be also saved.

The subjects who presented to ED Covid-19 outpatient clinic between March 11, 2020 and May 31, 2020 and for whom an infectious diseases (ID) physician was consulted (via Whatsapp or at bedside) will be included in the study in accordance with the inclusion and exclusion criteria.

In this cohort, the subjects whose consultations will be held before admission to another department, and the subjects inflicted with problems involving multiple departments were excluded from the study.In order to isolate potential Covid-19 patients during the pandemic process, these patients were examined at the Covid-19 outpatient clinic under the supervision of ED. Following their examination here, the consultation of those conforming to the potential Covid-19 patient classification will be held with ID department. The potential Covid-19 patients were assessed by an ED physician as specified in the Potential Covid-19 Cases Guide of Ministry of Health. In the Covid-19 pandemic period, not every consultation could be performed at bedside because both ED and ID physicians worked at a schedule twice as busy as normal times in relation to the congestion of working conditions and the organization of pandemic areas. During this pandemic process, consultations via Whatsapp emerged naturally due to the overcrowding in the pandemic outpatient clinic.

The eligible subjects examined by the ED physician who consulted an ID physician at the bedside or via Whatsapp will be evaluated in the study.

Whatsapp Consultation The ID physician was consulted for all the subjects once laboratory results and CT reports were complete. All the consultations were performed with the same smartphone, and every Whatsapp consultation held since the very beginning of the pandemic will be evaluated.

In this type of consultation, Thorax CT images of the patient were turned into a video of approximately 30-35 seconds, and during this video recording, the patient's clinical condition and laboratory results will be also transferred to the ID physician. The ID physician, on the other hand, stated his/her admission-discharge decision via Whatsapp as "hospitalization" or "discharge". Eventually the consultation result will be recorded in the patient's folder. The moment the video was sent will be recorded as the beginning of the patient's consultation period and response time to whatsapp video was saved as consultation response time.

The exclusion criteria in the present study can be listed as follows: the subjects whose consultations were held before admission to another department, the subjects inflicted with problems involving multiple departments and whose consultations were performed via Whatsapp, the subjects whose consultations were held by sending photos, the subjects who were referred from another outpatient clinic and whose consultation procedures were completed in ED and the subjects whose consultations were not replied on the same phone.

Since there is no reference study framed in a similar design, at least 90 people (45 people for each group) were needed to obtain 80% power with 95% confidence as a result of the power analysis conducted in line with the assumptions, presuming that the effect size we expected from the study would be high (f = 0.6).

The data will be analyzed with SPSS package program. Continuous variables were presented as median (IQR) while categorical variables will be provided as numbers and percentages. Kolmogrov-Smirnov analysis was used in normality distribution analysis. When the parametric assumptions were not met, the Mann-Whitney U test will be used to compare these differences. For all the analyses, P <0.05 will be considered statistically significant.

ELIGIBILITY:
Bedside consultation group

Inclusion Criteria:

.To be examined by the ED physician who consulted an ID physician only at the bedside.

Exclusion Criteria:

.To be consulted by the ED physician via whatsapp and at the bedside (both). .The patient's ID physician was consulted before completing the CT report and laboratory parameter results.

* The subjects whose consultations were held before admission to another department, .The subjects inflicted with problems involving multiple departments and whose consultations were performed via Whatsapp.
* The subjects who were referred from another outpatient clinic and whose consultation procedures were completed in ED

Whatsapp Consultation Inclusion Criteria To be consulted ID physician only only via whatsapp application. Exclusion Criteria

* The subjects whose consultations were held before admission to another department,
* The subjects inflicted with problems involving multiple departments and whose consultations were performed via Whatsapp,
* The subjects The subjects who were referred from another outpatient clinic and whose consultation procedures were completed in ED whose consultations were held by sending photos,
* The subjects who were referred from another outpatient clinic and whose consultation procedures were completed in ED .The subjects whose consultations were not replied on the same phone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The consultation method of the patients will be scanned retrospectively (from the fixed ED phone and the hospital system) and will be recorded in the dataset.
  Duration of video that send on whatsapp for consultation, infection diseases specialist response to video, clinician's response to bedside consultation will be saved to dataset. Besides, time from patients application to CT, time from patients application to lab results, duration of patients in ED and time periods of consultation (within working hour [8:00-17:00], or out of working hours [17:00-08:00]) will be also saved.
  The subjects who presented to ED Covid-19 outpatient clinic between March 11, 2020 and May 31, 2020 and for whom an infectious diseases (ID) physician was consulted (via Whatsapp or at bedside) were included in the study in accordance with the inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Analyzing the effect of consultation via whatsapp to lenght of stay the patients in emergency medicine department. | 1 month
  The effect of consultation via whatsapp to lenght of stay the patients in emergency medicine department will be analysed.

SECONDARY OUTCOMES:
Comparing the effect of bedside consultation and consultation via whatsapp on patient discharge or hospitalisation and readmission. | 1 month
  The effect of bedside consultation and consultation via whatsapp on patient discharge or hospitalisation and readmission will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Ramazan Sabirli, Kars, Outside of the US, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No planned to share.

REFERENCES:
- [Derived] Sabirli R, Karsli E, Canacik O, Ercin D, Ciftci H, Sahin L, Dolanbay T, Tutuncu EE. Use of WhatsApp for Polyclinic Consultation of Suspected Patients With COVID-19: Retrospective Case Control Study. JMIR Mhealth Uhealth. 2020 Dec 11;8(12):e22874. doi: 10.2196/22874. PMID 33276318